CLINICAL TRIAL: NCT02373553
Title: Impact of Physical Therapy Program in Mouthbreathing Children After Adenotonsillectomy: Randomized Clinical Trial.
Brief Title: Impact of Physical Therapy Program in Mouthbreathing Children After Adenotonsillectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, PATRICIA DAYRELL NEIVA, Master Degree in Rehabilitation Sciense, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3
Record Dates: First submitted 2015-02-23; First posted 2015-02-27 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Mouth Breathing
Keywords: posture; postural; kinetics
MeSH Terms: conditions — Mouth Breathing | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1( G1): CONTROL GROUP (No Intervention): not be submitted to intervention, only receive informations about health education.
- Group 2(G2) : HEALTH EDUCATION (Experimental): The family will receive a booklet of guidance of exercises to be performed at home.
  Interventions: Other: HEALTH EDUCATION
- Group 3(G3): EXERCISES IN OUTPATIENTS UNIT (Experimental): The postural reeducation through lengthening of the anterior muscles and strengthening of the posterior muscles of the trunk.
  Interventions: Other: EXERCISES

INTERVENTIONS:
Other: EXERCISES — The postural reeducation in a sitting position, in ventral and dorsal recumbency, including manual techniques, stretching the sternocleidomastoid and scalene muscles. Exercises for pelvic girdle positioning and stretching the hamstrings muscles tibial and sural triceps are associated with respiratory exercise. Twice a week during 3 months
  Arms: Group 3(G3): EXERCISES IN OUTPATIENTS UNIT
Other: HEALTH EDUCATION — Booklet contain many pictures demonstrating some exercises and an importance to do it.
  Arms: Group 2(G2) : HEALTH EDUCATION

SUMMARY:
MB Children maintains the same postural pattern in preoperative and postoperative adenotonsillectomy? The age influences the incidence of more exacerbated postural changes? The proposed early physiotherapy intervention can minimize future functional deficits? Trying to answer some of these questions, the objective of present study is to investigate the initial kinematics of the shoulder girdle, cervical and thoracic spine in MB children pre and post adenotonsillectomy and then evaluate the effects of a physical therapy intervention program for MB children who persisted with postural changes.

DETAILED DESCRIPTION:
Although oral breathing children be studied by otolaryngologists, allergists, orthodontists, speech therapists and physiotherapists and the prevalence of mouth breathing range from 26.6% to 53.3% in Brazilian studies, physical, medical and social problems arising from the Mouth Breathing Syndrome(MB) are still not recognized as a public health problem. Behavioral changes in sleep quality and craniofacial development and consequently the quality of life after surgical, orthodontic and multidisciplinary approach to the MB children are known.However, little is known about the effectiveness of early physical therapy intervention, whereas postural abnormalities characteristic of mouth breathing children are relevant and that the postural pattern adopted may persist into adulthood.

SPECIFIC OBJECTIVES

1. Compare linear measurements of elevation, scapular abduction and depression among MB children in preoperative and postoperative adenotonsillectomy.
2. Compare the angular measurements of upper / lower rotation, external / internal rotation, anterior / posterior tilt of the scapula and thoracic kyphosis, protrusion and retraction of the head and shoulders of protrusion and retraction group of MB children preoperative and postoperative adenotonsillectomy 3. Evaluate the impact of physical therapy intervention postoperatively.

STUDY DESIGN: Cohort cross-sectional PARTICIPANTS: The sample size calculation was based on the results of Correa et al (2008) , who report similar to the effects of intervention proposed in this study.45 children will be recruited from the Clinic of MOUTH BREATHING (ARO) of the Federal University of Minas Gerais (UFMG). To ensure adequate statistical power in case of loss to follow-up will be considered sample of 55 children.

ELIGIBILITY CRITERIA: 45 both male and female mouthbreathing children belonging to any racial group aged 4-10 years completed INCLUSION CRITERIA: diagnosis of upper airway obstruction by endoscopy (pharyngeal tonsil occupying 80% or more of the nasopharynx and / or palatine tonsils 3 or 4 ), history of oral route of access and loss of passive lip seal, display good understanding and whose family can signing the consent form approved by the Ethics Committee of the Federal University of Minas Gerais (COEP ).

EXCLUSION CRITERIA: children with neurological disorders, or endocrine abnormalities that compromise the normal development of growth, with the presence of ankylosis, severe lung disease, congenital heart defects, craniofacial abnormalities with syndromic and who are unfit to perform the procedures proposed in this study.

PROCEDURES Assessment and endoscopy will be held at ARO / UFMG where children will be screened according to the inclusion and exclusion criteria of this study. After passing the COEP, officials who accept to participate in the study must sign the Instrument of Consent. The collection of kinematic data will be held in the Motion Analysis Laboratory, Department of Physical Therapy. The physiotherapy intervention will be held at ARO, who works regularly on Thursdays for a period of three months.

STUDY PROTOCOL: Demographic and clinical data will be collected from all participants. All the measure proposed below will be obtained previously (T0) and three months after surgery (T1). By completing measures based process randomisation will be performed and the patients will be divided into 3 groups: GROUP 1(G1) - without physical interventions, only oral health education; GROUP 2 (G2)- guidance booklet for home with some stretched exercises and GROUP 3(G3) exercises -physiotherapy intervention proposal for a period of three months. After three months of allocation groups G1, G2 and G3 new measures will be carried out (T2). Those children who are identified with persistent postural changes will be forwarded to continue the specialized treatment.The G3 will be submitted to the postural reeducation through lengthening of the anterior muscles and strengthening of the posterior muscles of the trunk in a sitting position, in ventral and dorsal recumbency, including manual techniques, stretching the sternocleidomastoid and scalene muscles. Exercises for pelvic girdle positioning and stretching the hamstrings muscles tibial and sural triceps are associated with respiratory exercise. G2 family will receive a booklet of guidance of exercises to be performed at home and the G3 will not receive targeted intervention .

MEASURES: The kinematics of the shoulder girdle, cervical and thoracic spine of the participants will be obtained through the System Qualysis ProReflex ® in 3 times, regarding reliability. This is a photogrammetry system based on video that has four cameras with illumination stroboscopy produced by a group of infrared reflectors located around the lens of each camera. Infrared light designed for each camera is reflected by passive markers placed on specific points or anatomical points on the body of the participants. The reflection of light on passive markers is captured by cameras generating a two-dimensional (2D) image of the respective positions of these markers. The triangulation of the images of at least two cameras, allows the reconstruction in three dimensions (3D) passive reflective of brands. Data obtained are processed by the Track Manager software. Subsequently, data are transferred to the Mat Lab program (Matrix Laboratory) software, where the angular measurements are calculated using the arc tangent function. For the measurements of the orientation of the cervical spine, scapula, and thoracic spine, sixteen reflective tags are used, 15mm diameter.

TITLE:The orientation of the scapula includes three angular measurements (lower and upper rotation / anterior / posterior tilt, internal rotation / external) and two linear measurements (elevation and abduction). Upward rotation (U-Rot) A: occurs perpendicularly to the anterior-posterior axis and corresponds to the lateralization of the inferior angle of the scapula in relation to the spinal column on the frontal plane such that the glenoid cavity is oriented upwardly. Angle A was obtained from the intersection of a straight line passing through the C7 and T7 markers, a straight line passing through the medial edge of the scapula over the markers on the root of the spine and a marker over the inferior angle of the scapula.Scapular abduction (S-Abd) lateral shift of the scapula in relation to the spinal column. Horizontal distance (B) in millimeters from the centroid point of the scapula to the spinal column . Greater distance between markers indicated greater scapular abduction.Scapular elevation (S-Ele): linear upward shift of the scapular over the thoracic cage. C was obtained from the vertical distance in millimeters from the marker positioned over C7 to the centroid point of the scapula. Greater scapular elevation indicated a lesser distance between markers Measures of kyphosis of the thoracic spine, protraction / retraction and protraction of the head / shoulder retraction will also be undertaken.

TIME FRAME: 3 months after each assessment with safety issue INTERVENTION PROTOCOLS The G3 will be submitted to the postural reeducation through lengthening of the anterior muscles and strengthening of the posterior muscles of the trunk in a sitting position, in ventral and dorsal recumbency, including manual techniques, stretching the sternocleidomastoid and scalene muscles. Exercises for pelvic girdle positioning and stretching the hamstrings muscles tibial and sural triceps are associated with respiratory exercise. G2 family will receive a booklet of guidance of exercises to be performed at home and the G1 group did not receive intervention.

ELIGIBILITY:
Inclusion criteria: both sexes, belonging to any racial group aged 4-10 years completed, diagnosis of upper airway obstruction by endoscopy (pharyngeal tonsil occupying 80% or more of the nasopharynx and / or palatine tonsils 3 or 4 ), history of oral route of access and loss of passive lip seal, display good understanding and whose family can signing the consent form approved by the Ethics Committee of the Federal University of Minas Gerais (COEP ).

Exclusion criteria: children with neurological disorders, or endocrine abnormalities that compromise the normal development of growth, with the presence of ankylosis, severe lung disease, congenital heart defects, craniofacial abnormalities with syndromic and who are unfit to perform the procedures proposed in this study.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-02 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Angular and linear Measurement position of head, scapular and kyphosis | 1 year

SECONDARY OUTCOMES:
ages influences in this postural disorders | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia D Neiva, MD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] 1. Stokes, N. and Della, Mattia D. A student research review of the mouthbreathing habit: discussing measurement methods, manifestations and treatment of the mouthbreathing habit. Probe., v. 30, n. 6, p. 212-214, 1996. 2. Francesco, R. C., Passerotii, G., Paulucci, B., and Miniti, A. Respiração Oral na Criança:Repercussões diferentes de acordo com o diagnóstico. Rev.Bras.Otorrinolaringol., v. 70, n. 5, p. 665-670, 2004. 3. Aragao, W. Aragao's function regulator, the stomatognathic system and postural changes in children. J.Clin.Pediatr.Dent., v. 15, n. 4, p. 226-231, 1991. 4. Fujiki, P and R. Influência da hipertrofia adenoideana no crescimento e desenvolvimento craniodentofacial. Ortodontia, v. 32, n. 1, p. 70-77, 1999. 5.Lourenco, E. A. and Lopes, K. C. (1-2-2005). Estudo comparativo radiológico e nasofibroscópico do volume adenoideano em crianças respiradoras orais. Rev.Bras.Otorrinolaringol. 71[1], 23-28. 6. Lima, LCO, Baraúna, MA., Sologurem, MJJ, Canto, RST, and Gastaldi, AC. Postural alterations in children with mouth breathing assessed by computerized biophotogrammetry. J.Appl.Oral Sci., v. 12, n. 3, p. 232-237, 2004. 7. Krakauer, L. H. and Guilherme, A. Relationship between mouth breathing and postural alterations of children: a descriptive analysis. Int.J.Orofacial.Myology., v. 26, p. 13-23, 2000. 8. Yi, LC Pignatari S and Weckx LLM. Avaliação postural em crianças de 5 a 12 anos que apresentam respiração oral. Fisioterapia em movimento, v. 16, n. 3, p. 29-33, 2003. 9. Neiva PD, Kirkwood RN, Godinho R. Orientation and position of head posture, scapula and thoracic spine in mouth-breathing children. Int J Pediatr Otorhinolaryngol. 2009; 73:227-36.